CLINICAL TRIAL: NCT04105517
Title: Prescription of Hemangiol in the Treatment of Proliferative Infantile Hemangiomas Requiring Systemic Treatment: Post Marketing Surveillance Study
Brief Title: Hemangiol, Post Marketing Surveillance Study
Acronym: postHemangiol
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0402
Record Dates: First submitted 2019-09-18; First posted 2019-09-26 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Infantile Hemangioma
Keywords: Proliferative infantile hemangiomas; Hemangiol; Propranolol
MeSH Terms: conditions — Hemangioma, Capillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infantile hemangioma is a benign tumor belonging to the group of vascular tumors in the ISSVA classification (International Society for the Study of Vascular Anomalies). The diagnosis is clinical and radiological. The hemangioma appears during the first weeks of life (70% classically within 2 weeks after birth) but can, when it develops in the subcutaneous tissue, appear until the age of 2 to 3 months .

Its evolution is characteristic and is divided into 3 phases with a proliferative phase characterized by a rapid increase in the size of the tumor (up to 6 to 12 months), a phase of stabilization (from 12 to 36 months) with a stopping of the growth of the hemangioma and a regression of its size and a phase of involution with the disappearance of the lesion which may give way to residual fibroadipose tissue, cutaneous telangiectases, scars … The usual complications of haemangiomas occur during the proliferative phase. It is necrosis, ulcerations that can be complicated by bleeding or infection and eventually indelible scarring. Other complications related to the site of development of hemangiomas (amblyopia, astigmatism, upper respiratory obstruction, nasal obstruction, sphincter disorders, eating disorders), hemangiomas destroying structures noble (breast hypodévelopment, alopecia). The aesthetic prognosis can be seriously compromised for facial locations.

Historically, when drug therapy was required, patient management was based on systemic corticosteroids (at doses of 3 to 5 mg / kg / day) in first-line therapy and vincristine as a second-line failure of corticosteroid therapy or when life-threatening is at stake.

In 2014, the high French health authority (HAS) gave Marketing Authorization for Hemangiol 3.75 mg / ml oral solution for the management of infantile proliferative hemangioma requiring first-line systemic treatment, evaluating the actual benefit as important.

The selected indication concerns children from 5 weeks to 5 months with:

* Hemangiomas leading to a vital or functional risk,
* Hemangiomas ulcerated painful and / or not responding to simple care,
* Hemangiomas with a risk of permanent scarring or disfigurement. The 2014 HAS Transparency Commission wishes in its report "to have follow-up data of prescriptions allowing to describe on a representative sample of patients, the characteristics of the treated patients, the indication, the doses and the durations of treatment of this specialty ".

The objective of our study is to describe the use of Hemangiol in current practice in our hospital from 2014 to 2018.

DETAILED DESCRIPTION:
This study is retrospective, longitudinal, descriptive and observational. Children aged 0 to 1 years hospitalized for introduction of Hemangiol between January 2014 and November 2018 will be included. Patients refuse the use of medical data will be excluded.

The main objective is to describe the population who received Hemangiol. The secondary objectives is to evaluate

* the effectiveness of Hemangiol on proliferative infantile hemangiomas, -the tolerance of Hemangiol in children with proliferative infantile hemangiomas
* the interest of systematic cardiological consultation in children with proliferative infantile hemangiomas receiving Hemangiol

The following criteria will be collected

Demographic description: age, sex, height, weight

Personal history

Description of the hemangioma:

* organ concerned: skin, liver, parotid, mixed.
* location: head, thorax, pelvis, limbs, diffuse ...
* single or multiple
* indication of treatment: aesthetic, functional, ulcerated, cardiac hyperacidity

Rhythm of follow-up: duration of treatment and observance of treatment

Prescribed dose: 1, 2, 3 or 4 mg / kg / day in 2 doses

Evolution of the hemangioma: progression, regression, stagnation. Needed a second medical therapeutic line by specifying the treatment introduced. Necessity of surgical management by specifying the delay between surgery and the introduction of treatment

Description of serious adverse events: hypotension, bradycardia, bronchospasm, hypoglycaemia. Description of other adverse events.

Number of cardio-pediatric consultations, specifying:

* incidence of diagnosed heart disease through systematic cardiac consultation
* effect on ECG data of increasing dosage of Hemangiol: heart rate, PR duration, QRS duration, QT duration

ELIGIBILITY:
Inclusion criteria:

- Child from 0 to 18 years old hospitalized for introduction of Hemangiol between January 2014 and November 2018

Exclusion criteria:

- Patients refuse the use of medical data will be excluded.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 0 to 1 years hospitalized for introduction of Hemangiol for proliferative infantile hemangiomas.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events in children with proliferative infantile hemangiomas receiving Hemangiol | 6 days
  * rate serious adverse events: hypotension, bradycardia, bronchospasm, hypoglycemia
  * rate of adverse events

SECONDARY OUTCOMES:
Incidence of the regression of proliferative infantile hemangiomas in children receiving Hemangiol | 6 days
  rate of regression of the hemangioma
  * rate of need for a second therapeutic medical line
  * rate of need for surgical management
Incidence of diagnosed heart diseases with systematic cardiac consultation events in children with proliferative infantile hemangiomas receiving Hemangiol | 3 days
  rate of diagnosed heart disease

CONTACTS AND LOCATIONS:
Overall Officials: Arthur GAVOTTO, MD, Principal Investigator — University Hospital, Montpellier; Pascal AMEDRO, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Result] Socchi F, Bigorre M, Normandin M, Captier G, Bessis D, Mondain M, Blanchet C, Akkari M, Amedro P, Gavotto A. Hemangiol in infantile haemangioma: A paediatric post-marketing surveillance drug study. Br J Clin Pharmacol. 2021 Apr;87(4):1970-1980. doi: 10.1111/bcp.14593. Epub 2020 Nov 16. PMID 33118199